CLINICAL TRIAL: NCT07158970
Title: Effect of Home Ultrasound in Routine High-Risk Care of Patients With Gestational Diabetes Mellitus
Brief Title: Home-Ultrasound in Routine High-Risk Care of Patients With Gestational Diabetes Mellitus (GDM)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: PulseNmore (Industry)
Responsible Party: Principal Investigator, Liat Mor, OBGYN resident, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0125-25-WOMC
Record Dates: First submitted 2025-07-14; First posted 2025-09-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Gestational Diabetes Mellitus
Keywords: home ultrasound; telemedicine
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-US Group (Experimental): Home Ultrasound Monitoring
  Interventions: Device: Use of the Pulsenmore home ultrasound device for fetal assessment, guided remotely by a physician.
- Standard Care Group (No Intervention): Standard high-risk follow up in clinic

INTERVENTIONS:
Device: Use of the Pulsenmore home ultrasound device for fetal assessment, guided remotely by a physician. — Standard care
  Arms: Home-US Group

SUMMARY:
This study evaluates the impact of incorporating home-ultrasound (home-US) devices into telemedicine care for patients with gestational diabetes mellitus (GDM). The study will compare satisfaction, clinical outcomes, and healthcare costs between standard high-risk pregnancy care and care augmented by home-US.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) requires frequent follow-up to monitor maternal and fetal well-being. While telemedicine improves access and patient satisfaction, it lacks a fetal assessment component. This single-center randomized controlled trial evaluates the integration of home ultrasound (home-US) into telemedicine care for women with GDM.

Participants will be randomized to standard care or an intervention group receiving alternating in-person and telemedicine visits with physician-guided home-US using the Pulsenmore device. The primary outcome is patient satisfaction measured by the Diabetes Treatment Satisfaction Questionnaire (DTSQ) at term. Secondary outcomes include glycemic control, maternal and neonatal outcomes, healthcare utilization, visit duration, and follow-up costs.

The study will enroll 90 women, aged 18-51, with singleton pregnancies and GDM. The study is conducted at the Edith Wolfson Medical Center in Israel over a one-year period. The home-US device is approved for obstetric use and will be used under real-time physician supervision.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* GDM diagnosed by OGTT or glucose monitoring
* Hebrew speaking
* Compatible cellphone

Exclusion Criteria:

* Pregestational diabetes
* Fetal anomalies/genetic abnormalities
* Multifetal pregnancy
* Late GDM diagnosis (after 34 weeks)

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | at 37-39 weeks gestation
  Assessed using the Diabetes Treatment Satisfaction Questionnaire (DTSQ). It is composed of eight questions, each of which is scored by patients on a scale ranging from zero ("very dissatisfied", "very inconvenient") to six (e.g., "very satisfied", "very convenient").
  The questionnaire is composed of two different factors- the first 6 questions assess treatment satisfaction and the last 2 questions assess burden of hyper or hypo-glycemia. the sum of the first 6 points (maximum 36 points) score the treatment satisfaction, with a higher score indicating higher treatment satisfaction.

SECONDARY OUTCOMES:
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) Score | From enrollment (~24-28 weeks) to 37-39 weeks gestation.
  Difference in patient satisfaction as measured by the Diabetes Treatment Satisfaction Questionnaire (DTSQ) between early pregnancy (after first visit) and late pregnancy (37-39 weeks gestation).
  It is composed of eight questions, each of which is scored by patients on a scale ranging from zero ("very dissatisfied", "very inconvenient") to six (e.g., "very satisfied", "very convenient").
  The questionnaire is composed of two different factors- the first 6 questions assess treatment satisfaction and the last 2 questions assess burden of hyper or hypo-glycemia. the sum of the first 6 points (maximum 36 points) score the treatment satisfaction, with a higher score indicating higher treatment satisfaction.
Glycemic Control | From enrollment to delivery.
  Assessment of maternal glycemic control based on percent of abnormal glucose values during follow-up (via glucose log or continuous glucose monitoring where available), as recorded by treating physician.
Clinician Satisfaction | At the end of study participation for each patient (between 37-39 weeks gestation).
  Clinician satisfaction will be assessed using a structured questionnaire developed for this study. Physicians will rate various aspects of the telemedicine or in-person follow-up experience, including:
  Ease of use
  Clinical value
  Workflow and efficiency
  Communication and patient engagement
  Technical issues and support
  Each domain will be rated on a 10-point numeric rating scale (0-10), where:
  0 = Not satisfied at all
  10 = Extremely satisfied
  Higher scores indicate greater satisfaction.
Mode of Delivery | At time of delivery.
  Evaluation of mode of delivery (vaginal, cesarean)
Neonatal birth-weight | At time of delivery
  Birth weight
Estimated Patient Follow-up Costs | At 37-39 weeks gestation.
  Estimated costs incurred by patients for follow-up (including travel, parking, time off work), collected via structured questionnaire.
Estimated Institutional Follow-up Costs | From enrollment to delivery.
  Estimated resource and time costs for the healthcare system based on visit type (in-person vs. telemedicine), calculated per patient.
Visit Duration | Through study completion, an average of 1 year (from enrollment to delivery for each participant)
  Duration of each visit, separately recorded for patient time and physician Duration of each clinical visit will be recorded in minutes for both the patient and the physician. This includes both in-person and telemedicine encounters. Separate timing will be documented for:
  Patient time (including waiting and consultation)
  Physician time (active interaction and documentation)
  These data will be used to compare time efficiency between the two care models.
Unscheduled Emergency Department Visits | From enrollment to 6 weeks postpartum, confirmed by patient interview and EMR.
  Number and reason for unscheduled emergency room visits related to pregnancy or GDM during the study period.
Gestational age at birth | collected after birth from data system
  Gestational age at birth
Number of Neonates Admitted to the Neonatal Intensive Care Unit (NICU) | Within the first 28 days of life
  The number of neonates requiring admission to the neonatal intensive care unit (NICU) following delivery will be recorded and reported. This will be used as an indicator of neonatal morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: LIat Mor, Principal Investigator — Edith Wolfson Medical center
Locations (1):
- Edith Wolfson Medical Center, H̱olon, Central District, Israel

IPD SHARING:
Plan to Share IPD: No